CLINICAL TRIAL: NCT06268730
Title: Effects of SinuSonic on Psychological and Physical Well-Being In Adults With Nasal/Sinus Congestion
Brief Title: Effects of SinuSonic on Psychological and Physical Well-Being
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Healthy Humming LLC has ceased operating.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Healthy Humming, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-2437
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Nasal Congestion and Inflammations; Sinus Congestion Chronic
Keywords: anxiety; depression; autonomic reactivity; Polyvagal Theory; nasal congestion; adverse experience
MeSH Terms: conditions — Nasal Obstruction; Inflammation; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: All participants will follow the same procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SinuSonic (Experimental): Participants are asked to use the SinuSonic twice daily for 5 consecutive weeks. The duration of each use is 2 minutes.
  Interventions: Other: SinuSonic

INTERVENTIONS:
Other: SinuSonic — The SinuSonic is a commercially available, over-the-counter, self-applied nasal device designed to enhance physical well-being by reducing nasal congestion via simultaneous administration of acoustic vibration and gentle oscillating expiratory pressure.

SUMMARY:
The goal of this clinical trial is to evaluate the effects of using the SinuSonic on psychological and physical well-being in adults who have nasal/sinus congestion.

The study aims are:

* Aim #1: to evaluate the effect of the SinuSonic on physical and psychological well-being in individuals with chronic nasal congestion;
* Aim #2: to evaluate the relationship between autonomic reactivity and psychological well-being (i.e., anxiety and depression) in individuals with chronic nasal congestion;
* Exploratory Aim: to evaluate the impact of adverse experiences on physical and psychological well-being in individuals who experience chronic nasal congestion.

Participants will be asked to complete self-report measures of physical health, mental health and autonomic regulation before using SinuSonic (i.e., baseline research session) and after 5 weeks of directed use (post-intervention). Demographic information and adverse experiences will be documented during the baseline research session. Participants will be asked to document (weekly) current nasal symptoms and SinuSonic usage.

DETAILED DESCRIPTION:
All data collection will occur remotely using REDCap (via University of North Carolina, Chapel Hill) and SinuSonic use will take place in participants' homes. As this is a single-arm, feasibility/pilot study, all participants will follow the same protocol.

1. Baseline Research Session: self-report completion of demographic information, health information [Short Form Health Survey (SF-20), Total Nasal Symptom Score (TNSS)], autonomic reactivity (Body Perception Questionnaire, BPQ), anxiety/depression (Hospital Anxiety and Depression Scale, HADS), and adverse experiences (Adverse Traumatic Experiences Scale, ATES).
2. Begin use of SinuSonic twice per day, every day, for 5 weeks. Duration of each use is approximately 2 minutes. During these 5 weeks, participants will be asked to complete weekly forms to document SinuSonic usage and current nasal symptoms [Patient Global Impression of Change (PGIC), Total Nasal Symptom Score (TNSS).
3. Post-intervention Research Session: after 5 weeks of SinuSonic use, self-report completion of symptoms (PGIC, TNSS), autonomic reactivity (BPQ) and anxiety/depression (HADS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* US resident;
* Currently experiencing symptoms of nasal congestion that have persisted at least 2 weeks. Symptom severity must be rated at least 5, on a visual scale ranging from 1 to 10, as included in a question in the Eligibility Screening.

Exclusion Criteria:

* Previous use of the SinuSonic device.
* Meeting any of the conditions listed under the "Safety and Warnings" for using the SinuSonic device:

  1. Current or history of breathing problems (i.e., asthma, chronic obstructive pulmonary disorder (COPD), chronic bronchitis, emphysema, pneumonia, pleural effusion, lung cancer, cancer of the throat or upper airway)
  2. Current or history of circulatory problems (i.e., active nose bleed, heart arrhythmia, coronary artery disease, congestive heart failure, heart attack)
  3. Other conditions, specified as brain tumor, moderate to severe ear pain, fever greater than 101 degrees
  4. Pregnant or nursing women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keri J Heilman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months after publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 16 participants who signed informed consent and were enrolled, 4 did not complete any data collection or receive exposure to the study intervention. Twelve participants completed Baseline assessment.
Period: Overall Study
Arm/Group | SinuSonic
Started | 16
Completed Baseline | 12
Completed 5 Weeks | 7
Completed | 7
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | SinuSonic
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
  Chose not to answer | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Anxiety Subscale of the Hospital Anxiety and Depression Scale
Description: The Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of anxiety over the prior week. The anxiety subscale ranges from 0 to 21, with higher scores indicating higher anxiety complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Time Frame: Baseline, 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic
Number analyzed (Participants) | 7
score on a scale | -2.57 (1.24)
Statistical Analysis 1: Comparison: SinuSonic; Test type: Superiority; p = 0.104, ANOVA — The a priori threshold for statistical significance <0.05

2. Primary Outcome: Change in the Depression Subscale of the Hospital Anxiety and Depression Scale
Description: The Depression Subscale of the Hospital Anxiety and Depression Scale (HADS) is a 7-item self-report questionnaire measuring the frequency of depression over the prior week. The depression subscale ranges from 0 to 21, with higher scores indicating higher depression complaints. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Time Frame: Baseline, 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic
Number analyzed (Participants) | 7
score on a scale | -2.86 (1.25)
Statistical Analysis 1: Comparison: SinuSonic; Test type: Superiority; p = 0.061, ANOVA — the a priori threshold for statistical significance was <0.05

3. Secondary Outcome: Change in the Body Perception Questionnaire
Description: Body Perception Questionnaire (BPQ) is a self-report questionnaire, which includes a 20-item subscale for Autonomic Nervous System Reactivity. Only the Autonomic Nervous System Reactivity subscale will be administered. Raw scores range from 0-100, with higher scores indicating greater level of symptoms associated with autonomic activity (poorer outcome). Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Time Frame: Baseline, 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic
Number analyzed (Participants) | 7
score on a scale | -5.43 (2.49)
Statistical Analysis 1: Comparison: SinuSonic; Test type: Superiority; p = 0.053, ANOVA — the a priori threshold for statistical significance was <0.05

4. Secondary Outcome: Change in the Total Nasal Symptom Score
Description: Total Nasal Symptom Score (TNSS) is a 4-item self-report measure of congestion symptom severity. 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 12. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Time Frame: Baseline, 5 weeks
Population: Data are not reported for one participant who did not complete the initial questionaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic
Number analyzed (Participants) | 6
score on a scale | -3.67 (1.04)
Statistical Analysis 1: Comparison: SinuSonic; Test type: Superiority; p = 0.003, ANOVA — the a priori threshold for statistical significance was <0.05

5. Secondary Outcome: Change in the Patient Global Impression of Change
Description: The Patient Global Impression of Change (PGIC) is a 1-item self-report measure to rate the level of change that participants have experienced. The PGIC scale ranges from 1 to 7, with 1 indicating no change and 7 signifying a substantial improvement. Repeated measures ANOVA will be used to evaluate significant differences in change scores using a 0.05 significance level.
Time Frame: Week 1, Week 5
Population: Data are not reported for one participant who did not complete the Week 1 questionaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SinuSonic
Number analyzed (Participants) | 6
score on a scale | 0.50 (0.87)
Statistical Analysis 1: Comparison: SinuSonic; Test type: Superiority; p = 0.58, ANOVA — the a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Adverse Traumatic Experiences Survey at Baseline
Description: The Adverse Traumatic Experiences Survey (ATES) is a 30-item self-report measure with items relating to childhood adverse experiences, childhood maltreatment, other person maltreatment, life-threatening situations, sudden deaths of close ones, and personal health situations. Respondent-reported prior adverse events of maltreatment, life-threatening situations, and sudden deaths of close ones are summed to create an adversity score (range: 0-80), with higher scores indicating more adversity. Pearson correlational analysis will enable evaluation of the relationships between ATES and other Baseline outcome variables.
Time Frame: Baseline
Population: All collected data are reported although some participants opted not to complete all of the initial Baseline questionaires.
Measure: Number; unit: correlation coefficient
Arm/Group | SinuSonic
Number analyzed (Participants) | 11
correlation coefficient
  ATES with SF20: number analyzed (Participants) | 8
  ATES with SF20 | -0.39
  ATES with BPQ | 0.332
  ATES with HADS-Anxiety: number analyzed (Participants) | 10
  ATES with HADS-Anxiety | 0.543
  ATES with HADS-Depression | 0.492
  ATES with TNSS: number analyzed (Participants) | 10
  ATES with TNSS | -.002

7. Secondary Outcome: Short Form Health Survey (SF-20) at Baseline
Description: The 20-Item Short Form Survey (SF-20) is a shortened form of the original 36-item questionnaire created for the Medical Outcomes Study. The SF-20 utilizes close-ended, Likert-type questions to address self-reported health-related quality of life within six domains: physical functioning, role functioning, social functioning, mental health, current health perceptions, and pain. Raw scores from the 20 items are transformed linearly into 0-100 scales for each of the six domains. Higher scores indicate better physical, role, and social functioning, better mental health and health perceptions, and more pain. Scores across domains will be used to generate a general health status measure. Pearson correlational analysis will enable evaluation of the relationships between SF-20 and other Baseline outcome variables.
Time Frame: Baseline
Population: as for outcome 6
Measure: Number; unit: correlation coefficient
Arm/Group | SinuSonic
Number analyzed (Participants) | 9
correlation coefficient
  SF-20 with ATES: number analyzed (Participants) | 8
  SF-20 with ATES | -0.39
  SF-20 with BPQ | -0.66
  SF-20 with HADS-Anxiety: number analyzed (Participants) | 8
  SF-20 with HADS-Anxiety | -0.63
  SF-20 with HADS-Depression | -0.59
  SF-20 with TNSS | -.38

ADVERSE EVENTS:
Time Frame: From Baseline assessment through the end of study, up to 5 weeks.
Arm/Group | SinuSonic
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT06268730/Prot_SAP_000.pdf